CLINICAL TRIAL: NCT04619576
Title: Influence of the COVId-19 Pandemic on STRESS of Occupational Health Workers
Acronym: COVISTRESSWork
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 COVISTRESS Work
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Occupational Health
Keywords: COVID-19; Occupational health; Stress
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Occupational health workers — Questionnaire online

SUMMARY:
Coronavirus has caused containment of more than half of the world's population and a major and rapid reorganization of clinical and support services. The spread of coronavirus (COVID-19) has posed significant challenges for occupational health services. However, there is currently no data on the influence of this epidemic on the practice and feelings of dental surgeons and associates

DETAILED DESCRIPTION:
This is an observational study by REDCap questionnaire® via an internet link, which will be distributed to occupational health workers by any means The self-survey will assess stress, working conditions and changes in practices related to the coronavirus outbreak. This questionnaire includes 39 questions.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers who are screened

Exclusion Criteria:

* None

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Stress measures | Day 1
  Attitudes and stress related to screening procedure will be measured via questionnaire

SECONDARY OUTCOMES:
Sociodemographic characteristics | Day 1
  sociodemographic characteristics will be assessed by questionnaires
occupation perception | Day 1
  the perception about occupation will be assessed by questionnaires
work conditions | Day 1
  work conditions will be assessed by questionnaires
Changes in practices | Day 1
  changes in practices related to coronavirus pandemic will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, AURA, France